CLINICAL TRIAL: NCT03907618
Title: Evaluation of HbA1c Levels and Ovarian Reserve in Patients With Type 1 Diabetes Diagnosis
Brief Title: Evaluation of HbA1c Levels and Ovarian Reserve and Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, principal investigator, M.D, Department of Obstetrics and GynecologyR, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.10.22
Record Dates: First submitted 2019-04-06; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Diabetes; Ovarian Failure
Keywords: Antral follicle count; Anti müllerian hormone; Ovarian reserve; HbA1c; type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Ovarian Reserve

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 diagnosed with Diabetes Mellitus: Patients with Type 1 Diabetes Mellitus aged 18-40 years who had ovarian reserve with gynecological examination
  Interventions: Diagnostic Test: ovarian reserve
- group 2 control group: Healthy volunteer patients aged 18-40 years who have no diagnosis of Type 1 Diabetes Mellitus and whose ovarian reserve is evaluated by gynecological examination
  Interventions: Diagnostic Test: ovarian reserve

INTERVENTIONS:
Diagnostic Test: ovarian reserve — To assess ovarian reserve in patients with Type 1 Diabetes Mellitus aged 18-40 years; ultrasonographic and laboratory parameters will be looked at.

SUMMARY:
The human ovary is the target of an autoimmune attack, usually in organ or non-specific autoimmune disorders. Serum anti-Müllerian hormone (AMH) levels decrease early in menopause and menopause is seen in women with type 1 diabetes mellitus (DM1) at a young age. DM1 is aimed to show DM1 relationship with ovarian reserve based on the assumption that it will have lower AMH levels than controls, secondary to bad glycemic control and autoimmune attack in women.

DETAILED DESCRIPTION:
The study was designed prospectively. Ovarian functions in healthy volunteer women and patients who use DM1 diagnosed between 18-40 years old will be examined. Gonadotropin and AMH levels will be measured in follicular phase. To calculate the number of antral follicles (AFC) and ovarian volume, ultrasound will be looked at. Fasting and satiety blood glucose, HbA1c and C-peptide levels will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* female patients between 18 and 40 years of age who had consent and had gynecological examination in our polyclinic;
* study group for patients with type 1 diabetes mellitus healthy volunteers control group

Exclusion Criteria:

* Other endocrine and / or autoimmune disorders, polycystic ovary syndrome (PCOS) and
* previous surgery, which may reduce ovarian reserves;
* medical and / or radiotherapy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: female patients between 18 and 40 years of age who had consent and had gynecological examination in our polyclinic; study group for patients with type 1 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Antral follicle count (AFC) | On the 3rd day of the menstrual cycle
  AFC was calculated by counting 2-10 mm diameter follicles in both ovaries with a standard systematic approach.Recorded as a number.
Anti müllerian hormone (AMH) | On the 3rd day of the menstrual cycle
  AMH concentrations were measured by an enzymatically enhanced bilaterally immunoassay. AMH (pmol / l) saved as.
HbA1c | On the 3rd day of the menstrual cycle
  HBA1C concentrations were measured by taking venous blood samples in the early morning hours.
  HBA1C (mmol / mol) saved as.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)